CLINICAL TRIAL: NCT04600557
Title: A Compassion-based Intervention for Internal and External Shame
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor of Psychology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-07-0058
Record Dates: First submitted 2020-10-10; First posted 2020-10-23 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Shame; Compassion
Keywords: compassion; self-compassion; shame

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of four conditions throughout the study.
Who Masked: Participant
Masking Description: Participants are not told which arm they are assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-compassion only (Experimental): Describing a shameful experience using a self-compassionate prompt and receiving no verbal responses from confederates
  Interventions: Behavioral: Describing a shameful experience using a self-compassionate prompt; Behavioral: Receiving no response from confederates
- Compassion from others only (Experimental): Describing a shameful experience using a neutral prompt and receiving compassionate responses from confederates
  Interventions: Behavioral: Receiving compassionate responses from confederates; Behavioral: Describing a shameful experience using a neutral prompt
- Self-compassion plus compassion from others (Experimental): Both describing a shameful experience using a self-compassionate prompt and receiving compassionate responses from confederates
  Interventions: Behavioral: Describing a shameful experience using a self-compassionate prompt; Behavioral: Receiving compassionate responses from confederates
- Sharing-only control (Active Comparator): Describing a shameful experience using a neutral prompt and receiving no verbal responses from confederates
  Interventions: Behavioral: Describing a shameful experience using a neutral prompt; Behavioral: Receiving no response from confederates

INTERVENTIONS:
Behavioral: Describing a shameful experience using a self-compassionate prompt — Participants will be instructed to describe a shameful experience to two confederates using a self-compassionate prompt
  Other Names: Self-compassionate prompt
  Arms: Self-compassion only; Self-compassion plus compassion from others
Behavioral: Receiving compassionate responses from confederates — Following the participant's description of a shameful experience, two confederates will respond with compassionate responses
  Other Names: Compassionate confederates
  Arms: Compassion from others only; Self-compassion plus compassion from others
Behavioral: Describing a shameful experience using a neutral prompt — Participants will be instructed to describe a shameful experience to two confederates using a neutral (i.e., not self-compassionate) prompt
  Other Names: Neutral prompt
  Arms: Compassion from others only; Sharing-only control
Behavioral: Receiving no response from confederates — Following the participant's description of a shameful experience, two confederates will not be allowed to provide any verbal response
  Other Names: Neutral confederates
  Arms: Self-compassion only; Sharing-only control

SUMMARY:
This is a four-arm randomized pilot study aimed at reducing internal and/or external shame using self-compassion and/or compassion from others. The study is designed to test the theory that trait shame is comprised of both internal and external shame and to test compassion for others as an intervention for external shame.

DETAILED DESCRIPTION:
Shame is a common, painful emotion involving negative evaluations of the self. It has been theorized that trait shame involves both internal shame (i.e., evaluating oneself negatively) and external shame (i.e., perceiving that others evaluate the self negatively). Shame is experienced across a variety of psychiatric illnesses, yet it has been highly understudied.

Self-compassion has been used as an intervention for reducing shame in a variety of research studies, often in the context of a specific psychiatric disorder. However, self-compassion interventions, which aim to change the way one thinks and feels about oneself, may specifically target internal shame but not external shame. It is proposed that receiving compassion from others is an analogous and plausible intervention for external shame. In order to test the theory that trait shame is comprised of both internal and external shame and to test compassion for others as an intervention for external shame, a four-arm randomized pilot study aimed at reducing internal and/or external shame using self-compassion and/or compassion from others is proposed here.

Participants (N=180) scoring high on both internal and external shame on self-report measures will be assessed at baseline using both questionnaires and a shame-memory recall. Participants will be randomized to one of four conditions: a) describing a shameful experience using a self-compassionate prompt and receiving no verbal responses from confederates (self-compassion only), b) describing a shameful experience using a neutral prompt and receiving compassionate responses from confederates (compassion from others only), c) both describing a shameful experience using a self-compassionate prompt and receiving compassionate responses from confederates (self-compassion plus compassion from others), or d) describing a shameful experience using a neutral prompt and receiving no verbal responses from confederates (sharing-only control). Participants will complete questionnaires and shame-memory recalls again immediately following the sharing intervention and at a one-week post-intervention follow-up.

The two primary outcome measures will be state internal shame, as measured by the Internalized Shame Sclae, and state external shame, as measured by the Other As a Shamer scale. Both the Internalized Shame Scale and Other As a Shamer scale will be administered at baseline (immediately pre-treatment), immediately post-treatment, and a one-week post-intervention follow-up. Secondary outcome measures will include the Positive and Negative Affect Scale, and a real-time assessment of state shame.

It is expected that (a) participants assigned to describe a shameful experience using self-compassionate instructions will display larger reductions in internal shame relative to those assigned to describe a shameful experience using neutral instructions; (b) participants who receive compassionate responses from others after sharing a shameful experience will display larger reductions in external shame relative to those assigned to a listening-only control; and (c) participants assigned to describe a shameful experience using self-compassionate instructions combined with receiving compassionate responses from others will display larger reductions in both internal and external shame relative to participants who receive either component alone.

ELIGIBILITY:
Inclusion Criteria:

* Elevated levels of internal and external shame
* Can recall two shameful experiences

Exclusion Criteria:

* Active suicidal ideation as measured by endorsement of 2 (I would like to kill myself) or 3 (I would kill myself if I had the chance) on BDI-II item 9
* Endorses intent to harm or kill others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Internal shame | One-week post-intervention
  Measured by scores on Internalized Shame Scale (range: 0-120, higher indicates more shame)
Internal shame | 5 minutes post-intervention
  Measured by scores on Internalized Shame Scale (range: 0-120, higher indicates more shame)
External shame | One-week post-intervention
  Measured by scores on Other As Shamer Scale (range: 0-72, higher indicates more shame)
External shame | 5 minutes post-intervention
  Measured by scores on Other As Shamer Scale (range: 0-72, higher indicates more shame)

SECONDARY OUTCOMES:
Shame activation | 5 minutes post-intervention
  Real-time assessment of shame activation during shame memory recall tasks (range: 0-100)
Shame activation | one-week follow-up
  Real-time assessment of shame activation during shame memory recall tasks (range: 0-100)
State shame | 5 minutes post-intervention
  Micro-assessment of state shame using Positive and Negative Affect Scale (range: 1-5, higher indicates more shame)
State shame | one-week follow-up
  Micro-assessment of state shame using Positive and Negative Affect Scale (range: 1-5, higher indicates more shame)
Electrodermal response to shame | 5 minutes post-intervention
  Measured in microsiemens (μS) by Empatica E4 during shame memory recall tasks
Electrodermal response to shame | one-week follow-up
  Measured in microsiemens (μS) by Empatica E4 during shame memory recall tasks
Blood volume pulse in reaction to shame | 5 minutes post-intervention
  Changes in blood volume measured by Empatica E4 during shame memory recall tasks
Blood volume pulse in reaction to shame | one-week follow-up
  Changes in blood volume measured by Empatica E4 during shame memory recall tasks
Motion in reaction to shame | 5 minutes post-intervention
  Measured by 3-axis accelerometer sensor in the range [-2g, 2g] using Empatica E4 during shame memory recall tasks
Motion in reaction to shame | one-week follow-up
  Measured by 3-axis accelerometer sensor in the range [-2g, 2g] using Empatica E4 during shame memory recall tasks
Skin temperature reaction to shame | 5 minutes post-intervention
  Temperature measured in degrees Celcius by Empatica E4 during shame memory recall tasks
Skin temperature reaction to shame | one-week follow-up
  Temperature measured in degrees Celcius by Empatica E4 during shame memory recall tasks

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, PhD, Principal Investigator — Professor of Psychology
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook, D. R. Measuring shame: the internalized shame scale. Alcoholism Treatment Quarterly, 1987; 4, 197- 215.
- [Background] del Rosario, P.M., & White, R.M. The Internalized Shame Scale: Temporal stability, internal consistency, and principal components analysis. Personality and Individual Differences. 2006; 41, 95-103.
- [Background] Goss, K., Gilbert, P., & Allen, S. An exploration of shame measures-I: The Other As Shamer scale. Person. Individ. Diff.,1994; 17(5), 713-717.
- [Background] Andrews B, Qian M, Valentine JD. Predicting depressive symptoms with a new measure of shame: The Experience of Shame Scale. Br J Clin Psychol. 2002 Mar;41(Pt 1):29-42. doi: 10.1348/014466502163778. PMID 11931676
- [Background] Neff, K.D. The development and validation of a scale to measure self-compassion. Self and Identity. 2003; 2, 223-250.
- [Background] Rybak, C.J. & Brown, B. Assessment of internalized shame: Validity and reliability of the Internalized Shame Scale. Alcoholism Treatment Quarterly. 1996; 14:1.
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th ed.). Arlington, VA: American Psychiatric Publishing. 2013.
- [Background] Au TM, Sauer-Zavala S, King MW, Petrocchi N, Barlow DH, Litz BT. Compassion-Based Therapy for Trauma-Related Shame and Posttraumatic Stress: Initial Evaluation Using a Multiple Baseline Design. Behav Ther. 2017 Mar;48(2):207-221. doi: 10.1016/j.beth.2016.11.012. Epub 2016 Nov 29. PMID 28270331
- [Background] Gilbert P. The evolution of social attractiveness and its role in shame, humiliation, guilt and therapy. Br J Med Psychol. 1997 Jun;70(2):113-47. doi: 10.1111/j.2044-8341.1997.tb01893.x. PMID 9210990
- [Background] Gilbert, P. What Is shame? Some core issues and controversies. In Shame: Interpersonal behavior, psychopathology, and culture. 1998.
- [Background] Gilbert, P., & Procter, S. Compassionate mind training for people with high shame and self-criticism: Overview and pilot study of a group therapy approach. In Clinical Psychology and Psychotherapy. 2006; 13(6): 353-379. https://doi.org/10.1002/cpp.507
- [Background] Johnson, E. A., & O'Brien, K. A. Self-Compassion Soothes the Savage EGO-Threat System: Effects on Negative Affect, Shame, Rumination, and Depressive Symptoms. Journal of Social and Clinical Psychology. 2013; 32(9), 939-963. https://doi.org/10.1521/jscp.2013.32.9.939
- [Background] Judge, L., Cleghorn, A., McEwan, K., & Gilbert, P. An exploration of group-based compassion focused therapy for a heterogeneous range of clients presenting to a community mental health team. International Journal of Cognitive Therapy. 2012. https://doi.org/10.1521/ijct.2012.5.4.420
- [Background] Kim S, Thibodeau R, Jorgensen RS. Shame, guilt, and depressive symptoms: a meta-analytic review. Psychol Bull. 2011 Jan;137(1):68-96. doi: 10.1037/a0021466. PMID 21219057
- [Background] Lewis, M. Shame: The exposed self. New York: Free Press. 1992.
- [Background] Lewis, M. The role of the self in shame. Social Research, 70, 1181-1204. 2003.
- [Background] Luoma JB, Kohlenberg BS, Hayes SC, Fletcher L. Slow and steady wins the race: a randomized clinical trial of acceptance and commitment therapy targeting shame in substance use disorders. J Consult Clin Psychol. 2012 Feb;80(1):43-53. doi: 10.1037/a0026070. Epub 2011 Oct 31. PMID 22040285
- [Background] Skinta, M. D., Lezama, M., Wells, G., & Dilley, J. W. Acceptance and Compassion-Based Group Therapy to Reduce HIV Stigma. Cognitive and Behavioral Practice. 2015. https://doi.org/10.1016/j.cbpra.2014.05.006